

The Functional Gut Clinic 9<sup>th</sup> Floor, The Pinnacle 73-79 King Street Manchester M2 4NG

Phone: + 44 (0)161 302 7777

Email: enquiries@thefunctionalgutclinic.com

| <b>CONSENT FORM</b> | (Participant No:) |
|---------------------|-------------------|
|---------------------|-------------------|

Title of Project: The effect of an intestinal adsorbent on hydrogen and methane breath testing, in patients with abdominal and reflux symptoms, on long term proton pump inhibitor therapy

Name of Researcher: Dr Anthony Hobson

| | Please initial b | |
|---|---|---|
| 1. | I confirm that I have read and understand the information sheet dated 15/05/2019 (Version 3) for the above study. I have had the opportunity to consider the information, ask questions and have these answered satisfactorily. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | |
| 3. | I understand that relevant information on my medical history will be recorded and may be assessed by responsible individuals from the Chief Investigator's staff, FW medical or from the regulatory authorities, where it is relevant for regulatory purposes or in the case of an adverse event. I give permission for these individuals to have access to my study records. | , |
| 4. | I agree / do not agree (please circle as appropriate) that the study research team may inform my GP about my participation in the above named study. | |

| 5. | I would like to be informed of the results of the study once it has been completed | | | |
|---|---|---|---|---|
| 6. | I agree to take part in the above | e study. | | |
| <del></del><br>Na | me of Participant | Date | Signature | - |
| <br>Na | me of researcher taking consent | Date | Signature | - |

When completed 1 for participant; 1 for researcher site file; 1 (original) to be kept in participant notes.

# **Preflight Results**

### **Document Overview**

## Preflight Information

Title: Patient Identification Number for this trial: Profile: Convert to PDF/A-1b

**SMUHNT** Version: Author: Qoppa jPDFPreflight v2020R1.03

Microsoft® Word for Office 365 Jul 27, 2020 3:58:24 AM Creator: Date:

Producer: Microsoft® Word for Office 365

Legend: (X) - Can NOT be fixed by PDF/A-1b conversion.

(!X) - Could be fixed by PDF/A-1b conversion. User chose to be warned in PDF/A settings.

#### Page 1 Results

- (X) Font TimesNewRomanPSMT is not embedded.
- (X) Font TimesNewRomanPS-BoldMT is not embedded.
- (X) Font Arial-BoldMT is not embedded.
- (X) Font Arial-BoldMT is not embedded.
- (X) Font TimesNewRomanPS-BoldMT is not embedded.
- (X) Font TimesNewRomanPS-BoldMT is not embedded.
- (X) Font TimesNewRomanPS-BoldMT is not embedded.
- (X) Font ArialMT is not embedded.
- (X) Font ArialMT is not embedded.
- (X) Font ArialMT is not embedded.
- (X) Font TimesNewRomanPS-BoldMT is not embedded.
- (X) Font TimesNewRomanPS-BoldMT is not embedded.
- (X) Font TimesNewRomanPS-BoldMT is not embedded.
- (X) Font TimesNewRomanPSMT is not embedded. 102 more not displayed

#### Page 2 Results

- (X) Font TimesNewRomanPSMT is not embedded.
- (X) Font TimesNewRomanPSMT is not embedded.

#### Page 2 Results (contd.)

- (X) Font TimesNewRomanPSMT is not embedded.
- (X) Font TimesNewRomanPSMT is not embedded. 53 more not displayed